CLINICAL TRIAL: NCT01242618
Title: Tissue Engineered Nasal Cartilage for Reconstruction of the Alar Lobule Following Resection of a Non Melanoma Skin Cancer- a Phase I Clinical Trial.
Brief Title: Tissue Engineered Nasal Cartilage for Reconstruction of the Alar Lobule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TpP-I-2010-002
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Skin Carcinoma
Keywords: nasal cartilage diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- engineered nasal cartilage graft (Experimental): Biological intervention: autologous nasal chondrocytes expanded in vitro and cultured in a collagen Type I/III scaffold
  Interventions: Biological: engineered nasal cartilage graft

INTERVENTIONS:
Biological: engineered nasal cartilage graft — implantation of engineered nasal cartilage grafts in the alar lobule

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of implanting an engineered cartilage graft, obtained by culturing expanded autologous nasal chondrocytes within a collagen type I/III membrane, in the alar lobule of patients after resection of a non melanoma skin cancer.

DETAILED DESCRIPTION:
Skin cancer is the most prevalent reason for surgically creating a multilayer defect, consisting of skin and cartilage, of the alar lobule of the nose. In reconstruction of these defects, a combination of local flaps and autologous cartilage, typically harvested from the nasal septum or the ear, is used to restore the stability, function and proper 3D shape of the alar lobule. Harvesting autologous cartilage from the ear has been associated with a number of complications that could be overcome by the use of engineered cartilage graft generated in vitro with autologous cells.

This study is a phase I, prospective, uncontrolled, investigator initiated clinical trial involving 5 patients, with the objective of demonstrating safety and feasibility in the use of engineered nasal cartilage grafts. The specific surgical target of the trial is the reconstruction of a two layer defect of the alar lobule using a tissue engineered nasal cartilage graft and a local flap, following resection of a non melanoma skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* size of defect: ≥50% of alar subunit
* Extent of defect: 2 layer defect: skin and fibro-cartilaginous tissues

Exclusion Criteria:

* Defect extent:3 layers defect, including mucosa
* defect extent: 1 layer defect
* pregnancy
* immunodeficiency HIV
* Hepatitis B, C
* Allergy to porcine collagen, penicillin or streptomycin
* Chronic treatment with steroids or growth factors (immunomodulatory drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
safety: post operative complications should not be at higher rate than gold standard operative procedure. | 12 months post reconstruction
  Post operative complications could be: infections, bleeding, formation of scar tissue, asymmetry of the nostril to the opposite side

SECONDARY OUTCOMES:
feasibility of treatment | 12 months post reconstruction
  Functional testing of breathing Questionnaire of evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Martin, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Fulco I, Largo RD, Miot S, Wixmerten A, Martin I, Schaefer DJ, Haug MD. Toward clinical application of tissue-engineered cartilage. Facial Plast Surg. 2013 Apr;29(2):99-105. doi: 10.1055/s-0033-1341589. Epub 2013 Apr 5. PMID 23564241
- [Result] Fulco I, Miot S, Haug MD, Barbero A, Wixmerten A, Feliciano S, Wolf F, Jundt G, Marsano A, Farhadi J, Heberer M, Jakob M, Schaefer DJ, Martin I. Engineered autologous cartilage tissue for nasal reconstruction after tumour resection: an observational first-in-human trial. Lancet. 2014 Jul 26;384(9940):337-46. doi: 10.1016/S0140-6736(14)60544-4. Epub 2014 Apr 10. PMID 24726477